CLINICAL TRIAL: NCT02963454
Title: Effects of Levosimendan on Cellular Metabolic Alterations in Patients With Septic Shock: A Randomised Controlled Study
Brief Title: Effects of Levosimendan on Cellular Metabolic Alterations in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Hajjej Zied, Doctor, Military Hospital of Tunis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: LEVO02
Record Dates: First submitted 2016-11-04; First posted 2016-11-15 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Dobutamine; Simendan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- levosimendan 0.2 μg/kg/min (Experimental): Treatment with levosimendan 0.2 μg/kg/min 24h (without bolus).
  Muscle microdialysis was performed using a microdialysis probe inserted into the quadriceps femoris muscle.
  Interventions: Device: Microdialysis Probe (Muscle microdialysis); Drug: Levosimendan
- dobutamine 5 μg/kg/min (Active Comparator): Treatment with dobutamine 5 μg/kg/min. Dobutamine were administered during all the 72 hours study period.
  Muscle microdialysis was performed using a microdialysis probe inserted into the quadriceps femoris muscle.
  Interventions: Device: Microdialysis Probe (Muscle microdialysis); Drug: Dobutamine

INTERVENTIONS:
Device: Microdialysis Probe (Muscle microdialysis) — Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were determined at baseline and then every six hours for the following 72 hours after randomization.
  During the study period, conventional treatment was continued as per usual practice. Fluid challenges were performed, and repeated as necessary, to maintain central venous pressure (CVP) ≥8 and pulmonary arterial occlusion pressure (PAOP) ≥12 mmHg. Norepinephrine was titrated to maintain mean arterial pressure (MAP) ≥65 mmHg. Packed red blood cells were transfused when Hemoglobin (Hb) concentrations decreased below 7 g/dL, or if the patient exhibited clinical signs of inadequate systemic oxygen supply.
Drug: Dobutamine — Dobutamine (5 μg/kg/min) will be used as indicated
  Other Names: DOBUTREX
  Arms: dobutamine 5 μg/kg/min
Drug: Levosimendan — Levosimendan (0.2 μg/kg/min) will be used as indicated
  Other Names: SIMDAX
  Arms: levosimendan 0.2 μg/kg/min

SUMMARY:
To investigate changes in the concentration of glucose, lactate, pyruvate and glycerol in the extracellular fluid of the skeletal muscle following levosimendan administration in patients with septic shock.

DETAILED DESCRIPTION:
The study was designed as a prospective, double-blind, controlled, clinical trial and performed in a multidisciplinary intensive care unit. After achieving normovolemia and a mean arterial pressure of at least 65 mmHg, 20 septic shock patients were randomized to receive either levosimendan 0.2 μg/kg/min, or dobutamine 5 μg/kg/min. Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained by using muscle microdialysis. All measurements, including data from right heart catheterization were obtained at baseline and every 6 hours for the following 72 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

* patients who fulfilled the criteria of septic shock that required norepinephrine (NE) to maintain a mean arterial pressure (MAP) of at least 65 mm Hg despite appropriate volume resuscitation (pulmonary arterial occlusion pressure [PAOP] = 12 to 18 mm Hg and central venous pressure [CVP] = 8 to 12 mm Hg)

Exclusion Criteria:

* pregnancy, uncontrolled hemorrhage, terminal heart failure, significant valvular heart disease, documented or suspected acute coronary syndrome, and a limitation on the use of inotropes: left ventricle outflow obstruction, systolic anterior motion of the mitral valve.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
changes in the concentration of glucose(mmol/l) in the extracellular fluid of the skeletal muscle | At baseline and then every six hours for the following 72 hours after randomization.
changes in the concentration of lactate(mmol/l) in the extracellular fluid of the skeletal muscle | At baseline and then every six hours for the following 72 hours after randomization.
changes in the concentration of pyruvate (µmol/l) in the extracellular fluid of the skeletal muscle | At baseline and then every six hours for the following 72 hours after randomization.
changes in the concentration of glycerol (µmol/l) in the extracellular fluid of the skeletal muscle | At baseline and then every six hours for the following 72 hours after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: mustapha ferhjani, Study Director — Department of C ritical C are Medicine and Anesthesiology, Military Hospital of Tunis, Tunisia, Tunis, Tunisia
Locations (1):
- Military Hopital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No
via emails

REFERENCES:
- [Derived] Hajjej Z, Meddeb B, Sellami W, Labbene I, Morelli A, Ferjani M. Effects of Levosimendan on Cellular Metabolic Alterations in Patients With Septic Shock: A Randomized Controlled Pilot Study. Shock. 2017 Sep;48(3):307-312. doi: 10.1097/SHK.0000000000000851. PMID 28234790